CLINICAL TRIAL: NCT03793062
Title: Genetic and Epigenetic Basis of Chronic Wounds
Status: Recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Chandan Sen, Professor, University of Pittsburgh
Other Study IDs: STUDY23080025; R01DK135447 (NIH)
Record Dates: First submitted 2019-01-02; First posted 2019-01-04 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Chronic Wounds
Keywords: genome; epigenome; chronic wounds; genetics; socioeconomic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Wound debrided tissue, Blood, and Saliva samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No Interventions — Not applicable - No Interventions

SUMMARY:
This pilot study is designed for chronic wounds that fail to heal in a timely manner carry specific genetic signatures. These genetic signatures will be studied using debrided wound tissue that is removed by the wound care provider as part of standard of care. The reference genomic signature will be evaluated by obtaining blood samples and will be compared with wound debrided tissue genomic signature to understand wound specific genomic changes.

DETAILED DESCRIPTION:
Chronic wounds affect a large fraction of the world population and poses major threat to the public health and economy of the United States affecting 6.5 million patients. It has been estimated that approximately 2% of the population residing in developed countries, will experience at least one chronic wound during their lifetime. Current treatment options for chronic wounds are insufficient due to lack of individual specific genetic information. To improve therapy, an increase in the investigator's understanding of the genetic predisposition of individuals which result in impaired wound healing response is warranted. Information about these individual specific genetic and epigenetic regulations can altogether yield subset of repair genes which can serve as master regulators of wound healing. The effect of specific genetic information is also modified a lot by environmental epigenetic factors. Epigenetic changes have been shown to control the wound healing outcomes.

In this prospective pilot study, patients with chronic wounds visiting UPMC (University of Pittsburgh Medical Center) hospitals will be enrolled. Patients enrolled in the study will be followed for 16 weeks (+ or - 2 weeks). Within this time, debrided wound tissue will be collected, when available, as part of their standard of care at the clinics. The study consists of four study visits (Week 0, Week 4, Week 8 and Week 16 or earlier if target would is healed before that time). Study visit 1 consists of obtaining informed consent, medical history, current medications, and baseline demographics including, but not limited to: age, gender, zip code, ethnicity/race, marital status, education level, employment history, household income, number of household member. Digital imaging along with the collection of a saliva and blood sample will be performed during the visit. Participants will be asked to complete fourteen health questionnaires. Study visits two and three consists of digital imaging, along with a medication and adverse event review. Debridement tissue, if available, will be collected, if not collected earlier, during a follow up standard of care as part of wound care visit during the 16-week period. Study visit 4 (Healing Confirmation visit) consists of digital imaging, medication and adverse event review, along with Transepidermal water loss (TEWL) measurements.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Willing to comply with protocol instructions, including all study visits and study activities.
* Chronic wounds (> than four weeks since onset)
* Clinically diagnosed diabetic or non-diabetic ulcer.
* For patients with multiple wounds, the largest wound will be used for the study.

Exclusion Criteria:

* Individuals who are deemed unable to understand the procedures, risks and benefits of the study,(i.e. unable to provide informed consent)
* Pregnant females (self-declared) or lactating
* Subjects with marked immunodeficiency (HIV/AIDS or immune-suppressive medications)
* Prisoners

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 256 clinically diagnosed chronic wound patients will be recruited for this study.
Sampling Method: Non-Probability Sample
Enrollment: 256 (Estimated)
Dates: Start 2018-12-04 (Actual); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Epigenetic and transcriptome changes in debrided tissue from chronic wounds in healing vs non healing phase . | 16 weeks or healing whichever comes first
  The wound area (digital planimetry at d0/ 16 week) will classify wounds as heal-high (final 16 week size <40% of initial visit, d0) or heal-low (>60% of initial d0).
Wound specific genetic changes using whole genome approaches. | 16 weeks or healing whichever comes first
  To characterize wound specific genetic changes (e.g., mutations) using whole genome approaches. Genome from blood cells will be used as reference
Identify specific SEEBIN factors. | 16 weeks or healing whichever comes first
  To Determine the significance of socio-economic, environmental, behavioral, immunological and nutritional (SEEBIN) factors in modifying chronic wound (CW) tissue genomics in a way that affects healing trajectory.

CONTACTS AND LOCATIONS:
Overall Officials: Chandan K Sen, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Wound Care Centers, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Singer AJ, Clark RA. Cutaneous wound healing. N Engl J Med. 1999 Sep 2;341(10):738-46. doi: 10.1056/NEJM199909023411006. No abstract available. PMID 10471461
- [Background] Sen CK, Gordillo GM, Roy S, Kirsner R, Lambert L, Hunt TK, Gottrup F, Gurtner GC, Longaker MT. Human skin wounds: a major and snowballing threat to public health and the economy. Wound Repair Regen. 2009 Nov-Dec;17(6):763-71. doi: 10.1111/j.1524-475X.2009.00543.x. PMID 19903300
- [Background] Crovetti G, Martinelli G, Issi M, Barone M, Guizzardi M, Campanati B, Moroni M, Carabelli A. Platelet gel for healing cutaneous chronic wounds. Transfus Apher Sci. 2004 Apr;30(2):145-51. doi: 10.1016/j.transci.2004.01.004. PMID 15062754
- [Background] Gottrup F. A specialized wound-healing center concept: importance of a multidisciplinary department structure and surgical treatment facilities in the treatment of chronic wounds. Am J Surg. 2004 May;187(5A):38S-43S. doi: 10.1016/S0002-9610(03)00303-9. PMID 15147991
- [Background] Ti D, Li M, Fu X, Han W. Causes and consequences of epigenetic regulation in wound healing. Wound Repair Regen. 2014 May-Jun;22(3):305-12. doi: 10.1111/wrr.12160. PMID 24844330
- [Background] Mann J, Oakley F, Akiboye F, Elsharkawy A, Thorne AW, Mann DA. Regulation of myofibroblast transdifferentiation by DNA methylation and MeCP2: implications for wound healing and fibrogenesis. Cell Death Differ. 2007 Feb;14(2):275-85. doi: 10.1038/sj.cdd.4401979. Epub 2006 Jun 9. PMID 16763620
- [Background] Rahnama F, Shafiei F, Gluckman PD, Mitchell MD, Lobie PE. Epigenetic regulation of human trophoblastic cell migration and invasion. Endocrinology. 2006 Nov;147(11):5275-83. doi: 10.1210/en.2006-0288. Epub 2006 Aug 3. PMID 16887905
- [Background] Zhang W, Shiraishi A, Suzuki A, Zheng X, Kodama T, Ohashi Y. Expression and distribution of tissue transglutaminase in normal and injured rat cornea. Curr Eye Res. 2004 Jan;28(1):37-45. doi: 10.1076/ceyr.28.1.37.23493. PMID 14704912
- [Background] Ai L, Kim WJ, Demircan B, Dyer LM, Bray KJ, Skehan RR, Massoll NA, Brown KD. The transglutaminase 2 gene (TGM2), a potential molecular marker for chemotherapeutic drug sensitivity, is epigenetically silenced in breast cancer. Carcinogenesis. 2008 Mar;29(3):510-8. doi: 10.1093/carcin/bgm280. Epub 2008 Jan 3. PMID 18174247
- [Background] Chernov AV, Sounni NE, Remacle AG, Strongin AY. Epigenetic control of the invasion-promoting MT1-MMP/MMP-2/TIMP-2 axis in cancer cells. J Biol Chem. 2009 May 8;284(19):12727-34. doi: 10.1074/jbc.M900273200. Epub 2009 Mar 13. PMID 19286653